CLINICAL TRIAL: NCT05047666
Title: CLEAR: COVID-Like Illness Respiratory Pathogens - Diagnostics Response in Ghana. A Prospective Cohort on the COVID-19 Post-acute Condition
Brief Title: COVID-Like Illness Respiratory Pathogens. A Prospective Cohort on the COVID-19 Post-acute Condition
Acronym: CLEAR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Bernhard Nocht Institute for Tropical Medicine (Other Government)
Collaborators: Kumasi Centre for Collaborative Research (KCCR) (Other)
Responsible Party: Sponsor
Other Study IDs: CLEAR1.0
Record Dates: First submitted 2021-09-14; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Respiratory Infection; COVID-19 Respiratory Infection; Sequelae of; Infection
MeSH Terms: conditions — Respiratory Tract Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Respiratory samples (PCR), Blood Samples (Hematology, Biochemistry, Serology)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cases Group: Also called in our study 'Case-Positives'. These are those with respiratory symptoms suspected of COVID-19 that actually test positive (PCR).
- Symptomatic Control Group: Also called in our study 'Case-Negatives'. These are those with respiratory symptoms suspected of COVID-19 that actually test negative for SARS-CoV-2 but positive for any other pathogen included in our respiratory PCR-based panel.
- Healthy Control Group: At the community.

SUMMARY:
Identifying multiorgan sequalae and complications through high quality, prospective matched controlled studies throughout the course of COVID-19 is important for the acute and long-term management of patients and for health systems' planning. Further, it is key to understand the link between acute illness and long term consequences particularly in those already living with other comorbidities such as cardiovascular diseases or cancer.

Since the clinical presentation of COVID-19 can resemble a variety of common respiratory infections, describing the distribution of pathogens and the severity of clinical presentation associated with COVID-like illnesses (CLI) infections is important to generate a baseline clinical description by comparing potential long-term effects of PCR-confirmed COVID-19 to those following other respiratory infections.

To gain a better understanding of the clinical burden on COVID-19 survivors we will undertake a comparative evaluation within a cohort of PCR-confirmed individuals with COVID-19 vs. those PCR-confirmed symptomatic individuals with other respiratory pathogens plus healthy individuals from the community.

The results will inform strategies to prevent long term consequences; inform clinical management, interventional research, direct rehabilitation, and inform public health management to reduce overall morbidity and improve outcomes of COVID-19.

DETAILED DESCRIPTION:
This is an observational prospective matched cohort study to evaluate the post-acute consequences of the SARS-CoV-2 symptomatic infection (case-positives) while having as comparison groups (1) symptomatic controls (case-negatives) and (2) healthy controls, that are healthy individuals recruited from the same community of the cases, but not arise from the same household. After pre-screening of COVID-19 symptoms at the hospital and other satellite health centers, consenting/assenting patients of 16 years of age and above with all range of PCR-confirmed Covid-19 disease severity -from mild to severely ill hospitalized patients- will be recruited and matched to other Non-SARS-CoV-2 PCR-determined patients and to healthy community controls. Then, they will be followed up for 12 months (13 months after screening) to determine the occurrence of admissions, any outpatient encounter, symptoms (new or persistent) and concomitant use of medication after 28 days of diagnosis.

At recruitment, respiratory samples are collected for respiratory infections diagnosis. Also, blood samples are collected to generate baseline data on potential biomarkers associated to occurrence of investigated outcomes. This will include biochemistry (including inflammatory markers) and hematology as well as SARS-CoV-2 serology (IgG) which will also be taken at the end of follow up to rule out infection during the course of the follow up. Though, the serology testing won't be done along each recruitment but in batches during the study period. Clinical (symptoms and diagnosis), socioeconomic, demographic, household conditions, health seeking behavior and medical history information will be gathered.

ELIGIBILITY:
1. For symptomatic patients attending to the SFXH or other satellite health centers

   * Inclusion Criteria

     1. Patients > or =16 years of age
     2. Presenting respiratory symptoms
     3. Positive respiratory sample for SARS-CoV-2 or other respiratory infections included in the panel
     4. Possibility to be contacted during follow-up
     5. Consented participation
     6. Patients which households are located within the study catchment area
   * Exclusion Criteria

     1. Symptomatic patients who test negative for all pathogens of the PCR-based respiratory panel.
     2. Symptomatic patients who test negative for the SARS-CoV-2 RDT and do not meet the matching criteria (age and residency (community)) as symptomatic controls to any of the recruited cases (to be considered as controls for the Antimicrobial Use Workpackage)
2. Antimicrobial Use Work package (A subset of hospitalized, symptomatic patients are to be recruited as control group for the Antimicrobial Use Workpackage, if they meet the inclusion criteria)

   * Inclusion Criteria

     1. Patients > or =16 years of age
     2. Presenting respiratory symptoms
     3. Negative respiratory sample for SARS-CoV-2 (RDT)
     4. Do not meet the matching criteria (age and residency (community)) as symptomatic controls to any of the recruited cases
     5. Admitted to SFXH
     6. Consented participation
3. For healthy controls from the community

   * Inclusion Criteria

     1. Patients > or =16 years of age
     2. Meet the age and residency (community) criteria to be matched to the cases
     3. Possibility to be contacted during follow-up
     4. Consented participation
   * Exclusion Criteria

     1. Presenting COVID-19 like symptoms
     2. Positive for SARS-CoV-2 RDT Eligible participants in the community presenting with an acute illness can be considered for inclusion as a case and recommended for referral to SFXH/ satellite health centre.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study takes place in Assin Foso, Assin North District, Ghana. This is a semi rural area. Participants are recruited from the Saint Francis Xavier Hospital, the reference center of the region, when the seek for health services due to respiratory symptoms. Healthy controls are recruited from the communities from where cases arise.
Sampling Method: Non-Probability Sample
Enrollment: 1232 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Admissions and Outpatient encounter | 13 months
  Cumulated number of admissions and outpatient encounters within 13 months post PCR diagnosis
Persistent or new symptoms | 13 months
  Cumulated number of persistent/new symptoms within 13 months post PCR diagnosis
Medication and therapy | 13 months
  Cumulated therapy and use within 13 months post PCR diagnosis defined as:
  1. Average weekly intake of particular medication(s)
  2. Newly use of a particular medication(s)

SECONDARY OUTCOMES:
Patients' symptoms outcome | 13 months
  Occurrence of sequalae, post-acute symptoms and long-term patients' outcomes
Pathogen detection | 13 months
  Pathogens detected by PCR respiratory panel

OTHER OUTCOMES:
Exploratory Endpoint 1 | 13 months
  Viral variants detection via sequencing in the subgroup of symptomatic PCR-positive SARS-CoV-2 patients using the test-negative design.
Exploratory Endpoint 2 | 13 months
  Vaccine effectiveness in the subgroup of symptomatic PCR-positive SARS-CoV-2 patients using the test-negative design.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Strauss, Dr.MD. MPH, Principal Investigator — Bernhard Nocht Institute for Tropical Medicine; Jürgen May, Prof. Dr., Principal Investigator — Bernhard Nocht Institute for Tropical Medicine; Oumou Maiga-Ascofare, PhD, Principal Investigator — Kumasi Center for Collaborative Research in Tropical Medicine; John Amuasi, MBChB, MPH, PhD, Principal Investigator — Kumasi Center for Collaborative Research in Tropical Medicine